CLINICAL TRIAL: NCT03045822
Title: Evaluation of the Impact of Bioimpedance Analysis in Patients With Cardiac Implantable Electronic Devices
Brief Title: BIA and Cardiac Implantable Electronic Devices
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHU-302; 2013-A01060-45 (Other: 2013-A01060-45)
Record Dates: First submitted 2017-01-26; First posted 2017-02-08 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Performing Bioimpedance Analysis
Keywords: Bioimpedance analysis; implantable cardioverter-defibrillators; pacemakers

STUDY DESIGN:
Masking Description: open
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with cardiac implantable electronic devices (Experimental)
  Interventions: Drug: Bioimpedance analysis

INTERVENTIONS:
Drug: Bioimpedance analysis

SUMMARY:
There are an increase number of patients with cardiac implantable electronic devices (CIEDs) such as pacemakers (PM) and implantable cardioverter-defibrillators (ICDs) worldwide. The current medical practice guidelines warn on performing bioimpedance analysis (BIA) in this group of patients to avoid any electromagnetic interference. These recommendations restrict the use of BIA in many patients with heart failure in whom BIA might be of great interest in detecting peripheral congestion and in guidance of treatment. However, it is not well known whether BIA can affect the function of cardiac devices. Investigators aimed to test the incidence of electromagnetic interference between BIA and CIEDs.

DETAILED DESCRIPTION:
Patients enrollment were during routine face-to-face consultations, scheduled for PM and ICDs interrogations. Investigators recorded before and after each BIA measure, the battery voltage of the device, lead impedance and stimulation thresholds. The device electrograms were monitored during BIA measurements to detect any electromagnetic interference or oversensing.

ELIGIBILITY:
Inclusion Criteria:

* Patient having a cardiac device with or without cardiac resynchronization
* 18 years of age and above
* Patients with no pacing-dependent status
* Patients who read, understood and signed written informed consent letter

Exclusion Criteria:

* Patients with acute heart failure
* Patients implanted in less than 2 months
* Dysfunction of the device in a follow-up visit or in the inclusion visit
* Patients with a particular device lead model prone to develop electronical problems such as Sprint Fidelis of Medtronic (Minneapolis, USA) or Riata of St. Jude Medical (St. Paul, USA)
* Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-03-18 (Actual); Primary Completion 2016-02-28 (Actual); Study Completion 2017-01-16 (Actual)

PRIMARY OUTCOMES:
Assessing a change in CIEDs function while and after bioimpedance analysis | at 6 months

SECONDARY OUTCOMES:
Lead noise loss, over or under sensing of CIEDs | At 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric JEAN, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Chabin X, Taghli-Lamallem O, Mulliez A, Bordachar P, Jean F, Futier E, Massoullie G, Andonache M, Souteyrand G, Ploux S, Boirie Y, Richard R, Citron B, Lusson JR, Godet T, Pereira B, Motreff P, Clerfond G, Eschalier R. Bioimpedance analysis is safe in patients with implanted cardiac electronic devices. Clin Nutr. 2019 Apr;38(2):806-811. doi: 10.1016/j.clnu.2018.02.029. Epub 2018 Mar 2. PMID 29525512